CLINICAL TRIAL: NCT06287554
Title: Effect of Early Implementation of Prone Positioning Among Critically Ill Patients Admitted With Acute Respiratory Distress Syndrome During the COVID-19 Time: A Comparative Retrospective Observational Study
Brief Title: Effect of Early Implementation of Prone Positioning
Acronym: prone
Status: Completed | Type: Observational
Sponsor: Zulekha Hospitals (Other)
Collaborators: Al-Azhar University (Other)
Responsible Party: Sponsor
Other Study IDs: 404/2024
Record Dates: First submitted 2024-02-23; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Severe Acute Respiratory Syndrome
Keywords: Prone, Lung protective, ARDS, APACHI II, SOFA
MeSH Terms: conditions — Severe Acute Respiratory Syndrome | interventions — Prone Position

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 26 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Group A (n:39) included patients who had been early placed in prone positions within 24 hours of intubation
  Interventions: Other: PRONE POSITION
- Group B: Group B (n:31) included patients who had not been placed in prone position

INTERVENTIONS:
Other: PRONE POSITION — early placed in prone positions within 24 hours of intubation
  Groups: Group A

SUMMARY:
Background and objective: The ramifications of early lung protective measures and prone positioning on the ICU length of stay rates of participants admitted to the ICU with acute respiratory distress syndrome amid the COVID-19 pandemic constitute a pivotal examination. The study aims to identify the effect of early prone positioning on the length of stay, discharge rate, and number of tracheostomized patients in the ICU.

DETAILED DESCRIPTION:
Background and objective: The ramifications of early lung protective measures and prone positioning on the ICU length of stay rates of participants admitted to the ICU with acute respiratory distress syndrome amid the COVID-19 pandemic constitute a pivotal examination. The study aims to identify the effect of early prone positioning on the length of stay, discharge rate, and number of tracheostomized patients in the ICU.

Methodology: This retrospective study was conducted on critically ill patients needing mechanical ventilation with lung protective strategy and admitted to the Intensive Care Units of Al-Azhar University Hospitals between March 2020 to April 2022. All patients in the study were interpreted retrospectively by examining the patient's records. Group A (n:39) included patients who had been early placed in prone positions within 24 hours of intubation, and Group B (n:31) included patients who had not been placed in prone positions. All patients received a lung protective strategy for ARDS. In both groups, PaO2, PaCo2, PH, SpO2, and PaO2/FiO2 ratio were checked initially and later every 24 hours for 6 days. All patients were evaluated for the total days of both hospital and ICU length of stay, number of successful discharges to home from the hospital, and the total number of tracheostomized patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients of both sexes.
* Aged from 18 to 70 years.
* Body Mass Index (BMI) from 25 to 35 kg/m2.
* Critically ill due to ARDS resulting from COVID-19 pneumonia.

Exclusion Criteria:

* Patients who spent more than 24 hours on mechanical ventilators before enrolment in the study.
* Patients who died within the first 24 hours of presentation.
* Patients with advanced cancer.
* Pregnant patients.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 124 patients were recruited initially to the study who were admitted with ARDS to the ICU. A total of 70 patients were finally included and divided into two groups,
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2020-03-04 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
Number of discharged patients | 26 MONTHS
  Number of discharged patients

SECONDARY OUTCOMES:
The total length of stay | 26 MONTHS
  The total length of stay
ICU length of stay | 26 MONTHS
  ICU length of stay
Patients who underwent tracheostomy procedures | 26 MONTHS
  Patients who underwent tracheostomy procedures

CONTACTS AND LOCATIONS:
Overall Officials: SAMEH H SEYAM, PHD, Study Chair — Consultant critical care
Locations (1):
- Al-Azhar faculty of medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
undecided